CLINICAL TRIAL: NCT03033667
Title: Comparative Study Between Conventional Fasting Versus Overnight Infusion of Lipid or Carbohydrate on Free Fatty Acid and Insulin in Obese Patients Undergoing Elective First Time On-pump Coronary Artery Bypass Grafting
Brief Title: Conventional Fasting Versus Lipid/Carbohydrate Infusion for Coronary Bypass Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Hosny, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMOF
Record Dates: First submitted 2017-01-06; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Metabolism Disorder
Keywords: perioperative fasting; free fatty acids; coronary bypass grfting
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucose group (G group) (Experimental): patients received 500 cc of glucose 10% that containing 50 g of glucose and provides patients with 200 Kcal with 556 mosmoles/L.
  Interventions: Dietary Supplement: G group
- Lipid Group (L group) (Experimental): patients received 100 cc of lipid solution (soybean 30%, medium chain triglycerides 30%,olive oil 25%,fish oil 15% and 20 mg vitamine E) containing 20 g lipid and provides patients with 200 Kcal with osmolarity of 380 mosmoles /L.
  Interventions: Dietary Supplement: group L
- Control Group (C group) (Experimental): patients was fasting overnight from 11 pm till 9 am except for clear fluids that was allowed till 5 am.
  Interventions: Dietary Supplement: Group C

INTERVENTIONS:
Dietary Supplement: G group — patients received 500 cc of glucose 10% containing 50 g of glucose proving patients with 200 Kcal with 556 mosmoles/L
  Arms: Glucose group (G group)
Dietary Supplement: group L — patients received 100 cc of lipid solution (soybean 30%, medium chain triglycerides 30%,olive oil 25%,fish oil 15% and 20 mg vitamine E) containing 20 g lipid which provided patients with 200 Kcal with osmolarity of 380 mosmoles /L. with a flow rate of infusion of 12.5 cc per hour
  Arms: Lipid Group (L group)
Dietary Supplement: Group C — Over night fasting with no supplementation
  Arms: Control Group (C group)

SUMMARY:
Comparative study between conventional fasting versus overnight infusion of lipid or carbohydrate on free fatty acids and insulin in obese patients undergoing elective first time on-pump coronary artery bypass grafting.

DETAILED DESCRIPTION:
Obese patients scheduled for bypass surgery randomly assigned to three groups:

Group I (Glucose-group): patients received 500 cc of glucose 10% containing 50 g of glucose and providing patients with 200 Kcal with an osmolarity of 556 mosm/L.

Group II (Lipid-group): patients received 100 cc of lipid solution (soybean 30%, medium chain triglycerides 30%,olive oil 25%,fish oil 15% and 20 mg vitamine E) containing 20 g lipid and provides patients with 200 Kcal with an osmolarity of 380 mosm/L.

Group III (Control-group): patients fasted overnight from 11 pm till 9 am except for clear fluids which were allowed till 5 am.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (> 18 years) with American Society of Anesthesia (ASA) class II-III, BMI 30-40, and New York Heart Association (NYHA) functional capacities I-II, undergoing elective on-pump coronary artery bypass grafting (CABG) using cardiopulmonary bypass (CPB).

All patients were type 1a World Health Organisation (WHO)/Fredrickson classification of primary hyperlipidemias.

Exclusion Criteria:

* Patients with diabetes mellitus
* Patients on fibrates
* Patients type 1,2b,3,4 and 5 WHO/Fredrickson classification of primary hyperperlipidemias
* Patients with history of allergic reactions to fish, egg yolk containing foods peanut or soy products
* Patients with carbohydrate or fat intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The change in free fatty acids levels and insulin blood levels before and after the infusion of study solution | Over an infusion period of 10 hours preoperatively

IPD SHARING:
Plan to Share IPD: Yes